CLINICAL TRIAL: NCT00018850
Title: 5HT3 Antagonism and Auditory Gating in Schizophrenia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: MHBS-013-99F
Record Dates: First submitted 2001-07-03; First posted 2001-07-05 (Estimated); Last update posted 2009-01-21 (Estimated); Status verified 2004-12

CONDITIONS: Schizophrenia
Keywords: schizophrenia; ondansetron; nicotine; haloperidol
MeSH Terms: conditions — Schizophrenia | interventions — Ondansetron; Neuropsychological Tests; Nicotine; Haloperidol

INTERVENTIONS:
Drug: ondansetron
Behavioral: neuropsychological testing
Drug: nicotine
Drug: haloperidol

SUMMARY:
The target groups in this study are brain waves and neurotransmitters (chemical messengers) in the brain. Subjects with diagnosed with schizophrenia will be studied. The study will help understand more about normal brain functioning and how that functioning differs in people with schizophrenia. Another purpose of this study is to determine how the altered brain functioning in schizophrenia contributes the symptoms found in the illness.

ELIGIBILITY:
Subjects with diagnosed with schizophrenia will be studied.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Dates: Start 1998-06; Study Completion 2003-06

CONTACTS AND LOCATIONS:
Locations (1):
- VAMC, Denver, Colorado, United States